CLINICAL TRIAL: NCT03102476
Title: A Study to Assess Environmental Effects of Temperature and Humidity on Pharmacokinetics and Pharmacodynamics of Prandial Insulin in Subjects With Type 1 Diabetes
Brief Title: Environmental Effects Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Principal Investigator, Thozhukat Sathyapalan, Professor, University of Hull
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Version: 3.0 (02-07-2014)
Record Dates: First submitted 2016-12-06; First posted 2017-04-05 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2017-03

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Insulin Lispro

ARMS (1):
- Patients with Type 1 Diabetes (Other): Using euglycaemic clamp, the effect of different temperatures and humidity levels will be assessed on the pharmacokinetic and pharmacodynamic profiles of short-acting insulin Humalog.
  Interventions: Drug: Humalog

INTERVENTIONS:
Drug: Humalog — Subcutaneous injection of Humalog and assessing Pharmacokinetics and Pharmacodynamics properties of Humalog under different environmental conditions
  Other Names: Insulin lispro

SUMMARY:
Type 1 Diabetes mellitus (T1D) is characterized by βcell destruction and a long life requirement of exogenous insulin. The bolus basal insulin regimen is a widely accepted therapy concept to treat hyperglycaemia in patients with T1D. This concept requires a very good knowledge of the individuals prandial and basal insulin requirements. However, insulin requirement depends on insulin absorption from the injection site and the individual's insulin sensitivity which relies on a number of effects including body composition, inflammatory processes and environmental factors. Climatic factors such as differences in air temperature could affect both, insulin absorption and insulin sensitivity as suggested by recent reports. For instance, it is reported that hot baths can accelerate the absorption of short acting but not of long acting insulin formulations from the subcutaneous depot. In addition, local warming of the injection site by a novel device (InsuPatch) results as well in an accelerated insulin action profile of short acting insulins. Moreover, Berglund et al. reported seasonal variations in insulin sensitivity in elderly men with increased insulin sensitivity during summer time.

Although an effect of temperature on insulin absorption and action can be assumed and was subject to current clinical trials, there is only little knowledge on the effect of humidity and the cumulative effect of humidity and temperature on insulin pharmacodynamics and pharmacokinetics. For subjects with type 2 diabetes it was reported that accommodation to high temperatures and moist air of more than 75% is impaired compared to healthy subjects as determined by skin blood flow, temperature and moisture. Although it can be estimated that changes in blood flow due to hot and moist air affect the pharmacokinetics and pharmacodynamics of subcutaneous prandial insulins, to our knowledge no such study in subjects with T1D using the euglycaemic clamp technique was carried out yet. In order to assess the effect of temperature and humidity on insulin action, subjects with type 1 diabetes will be administered a single dose of short acting insulin in an environmental chamber either at 15°C or a warm environment of 40°C with either a low or high humidity (10% vs. 90%). Moreover, an exploratory part of the trial will evaluate the measurement performance of several blood glucose meters under the experimental climatic situations.

DETAILED DESCRIPTION:
BACKGROUND Type 1 Diabetes mellitus (T1DM) is characterised by β-cell destruction and a lifelong requirement of exogenous insulin. The basal-bolus insulin regimen is widely accepted therapy to treat hyperglycaemia in patients with T1DM. This concept requires a very good knowledge of the individual's prandial and basal insulin requirements. However, insulin requirement depends on insulin absorption from the injection site and the individual's insulin sensitivity that relies on a number of factors including body composition, inflammatory processes and environmental factors. Environmental factors such as differences in air temperature could affect both, insulin absorption and insulin sensitivity as suggested by recent reports. For instance, it is reported that hot baths can accelerate the absorption of short-acting but not of long-acting insulin formulations from the subcutaneous depot. In addition, local warming of the injection site by a novel device (InsuPatch) results in an accelerated insulin-action profile of short-acting insulins. Moreover, Berglund et al. reported seasonal variations in insulin sensitivity in elderly men with increased insulin sensitivity during summer time.

Although an effect of temperature on insulin absorption and action can be assumed, there is only little knowledge on the effect of humidity and the cumulative effect of humidity and temperature on insulin pharmacodynamics and pharmacokinetics. For subjects with type 2 diabetes it was reported that accommodation to high temperatures and moist air of more than 75% is impaired compared to healthy subjects as determined by skin blood flow, temperature and moisture.

Although it can be estimated that changes in blood flow due to hot and moist air affect the pharmacokinetics and pharmacodynamics of subcutaneous prandial insulins, to our knowledge no such study in subjects with T1D using the euglycaemic clamp technique has been performed. In order to assess the effect of temperature and humidity on insulin action, subjects with type 1 diabetes will be given a single dose of short-acting insulin in an environmental chamber either at 15°C or a warm environment of 30°C with either a low or high humidity (10% vs. 60%).

TRIAL OBJECTIVES The objective of this trial is to assess the effect of different temperatures and humidity levels on the pharmacokinetic and pharmacodynamic profiles of short-acting insulin in subjects with type 1 diabetes mellitus.

TRIAL DESIGN The trial will be a single-centre, open label, 3-way cross-over, euglycaemic glucose clamp trial in subjects with type 1 diabetes mellitus. The pharmacodynamic and pharmacokinetic properties of insulin Humalog dosed at 0.2 U/kg will be investigated.

ENVIRONMENTAL SETTINGS

* 15 °C and 10% humidity
* 30 °C and 10% humidity
* 30 °C and 60% humidity

ASSESSMENTS

* 6 visits to the clinical unit: informed consent and screening visit (Visit 1, within 28 days prior to Visit 2a), Pre-dosing visit (Visit 2a, within 3 days of 2b), 3 dosing visits (Visit 2b, 3 & 4, wash-out period of 3-21 days between each visit), and 1 follow-up (FUP) examination (Visit 5, 3-14 days after last dosing visit)
* Change in insulin regimen (72 hours prior to each dosing):

The patients will be switched from Insulin Lantus or detemir to NPH 48 hours before dosing visit. The NPH insulin will then be stopped 22 hours before dosing visit except short acting insulin which will be stopped 6-8 hours before visit.

* Euglycaemic clamp setting for 6 hours after administration on dosing Visits 2b, 3 & 4
* Blood to be collected for the determination of PK insulin concentrations on Visit 2b, 3 & 4 before and after administration of insulin
* Blood glucose will be continuously monitored pre-administration and for 6 hours after administration of insulin
* Determination of skin blood flow via Laser-Doppler
* Standard safety parameters will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Diabetes mellitus type 1
* HbA1c ≤ 9.0 %
* Total insulin dose of < 1.2 U/kg/day
* Age between 18 and 55 years, both inclusive
* Body mass index (BMI) between 18.0 and 28.0 kg/m2, both inclusive
* Informed consent must be obtained for all volunteers in writing

Exclusion Criteria:

* Known or suspected allergy to insulin.
* Recurrent major hypoglycaemia or hypoglycaemic unawareness as judged by the Investigator or hospitalization for diabetic ketoacidosis during the previous 6 months.
* Clinically significant diabetic neuropathy, in particular autonomous diabetic neuropathy.
* Supine blood pressure at screening (after resting for 5 min in supine position) outside the range of 90-140 mmHg for systolic or 50-90 mmHg for diastolic (excluding white-coat hypertension; therefore, if a repeated measurement shows values within the range, the subject can be included in the trial) and/or resting supine heart rate outside the range 50 -90 beats per minute. This exclusion criterion also pertains to subjects being on antihypertensives.
* Treatment with any other investigational drug within 3 months prior to screening. Participation in a clinical research trial in last 3 months.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve from 0 hours until the end of clamp. | 1 Year
Onset of action, time from trial product administration until the blood glucose concentration has decreased at least 0.3 mmol/L (5 mg/dL) from the baseline | I year

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve from 0 hours until 2 hours | 1 year
Area under the glucose infusion rate curve from 0 hours until 4 hours | 1 year
Area under the glucose infusion rate curve from 0 hours until 6 hours | 1 year
Area under the glucose infusion rate curve from 4 hours until 6 hours | 1 year
Maximum glucose infusion rate | 1 year
Time to maximum glucose infusion rate curve | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thozhukat Sathyapalan, MD FRCP, Principal Investigator — United Kingdom: Hull University
Locations (1):
- Hull and East Yorkshire NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided